CLINICAL TRIAL: NCT00025714
Title: Research Study of Specimens Obtained During Epilepsy Surgery
Brief Title: Study of Specimens Obtained During Epilepsy Surgery
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020014; 02-N-0014
Record Dates: First submitted 2001-10-11; First posted 2001-10-12 (Estimated); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy
Keywords: Serotonin Receptor; Cell Culture; Temporal Lobe; Endothelial Cells; Superficial Temporal Artery; Natural History; Epilepsy; Intractable Epilepsy
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients who have agreed to undergo brain surgery to treat drug resistant epilepsy and are enrolled in protocol 11-N-0051 Epilepsy Surgery.

SUMMARY:
This study will collect brain tissue samples for research purposes from patients undergoing surgery to treat epilepsy. The standard surgical procedure for medically intractable epilepsy i.e., epilepsy that cannot be controlled with medicine requires removal of more brain tissue than is needed for diagnostic study. This extra tissue, which would otherwise be discarded, will be used for research purposes. In addition, a blood vessel in the scalp, called the superficial temporal artery, is also normally cut during surgery, and a piece of this vessel will be taken for research use.

Patients 4 years of age or older who undergo surgery for medically intractable epilepsy may be eligible for this study.

Brain tissue collected under this protocol will be used for studies of brain cells in other diseases and of serotonin receptors. Any remaining brain tissue will be frozen for use in future research. The superficial temporal artery will be used for comparison with carotid arteries (a neck artery that supplies the brain) from patients with blockage of this blood vessel.

DETAILED DESCRIPTION:
This is a protocol to perform research studies on tissues that are removed in the operating room during surgical procedures for drug resistant epilepsy. Our aim is to acquire and supply useful tissue specimens for intramural NIH research projects.

The investigators will evaluate participants with medically intractable drug resistant epilepsy who are considered for surgery to determine whether surgical specimen may be available for this protocol. Surgery and standard care for these participants will be performed under a separate protocol, 11-N-0051 Epilepsy Surgery. The intent of this protocol is solely for procuring tissue that is resected for standard clinical care during surgery. This protocol is not designed to test any new treatments.

These are the research aspects of the protocol: 1) Any brain tissue that is removed and is not required for diagnostic studies will be used for laboratory studies, consistent with institutional guidelines. 2) Blood tests to test for immune and inflammatory mediators will be performed. 3) Saliva will be collected to test for immune and inflammatory markers.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for entry into the study, candidates must meet al the following criteria:

1. Be 4 years of age or older.
2. Able to give informed consent, or, assent if a child.
3. Have agreed to undergo brain surgery to treat drug resistant epilepsy and are enrolled in protocol 11-N-0051 Epilepsy Surgery.

EXCLUSION CRITERIA:

Candidates will be excluded if they:

1. Are not a surgical candidate as specified in appropriate protocols.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participant population for this study is restricted to participants with drug resistant epilepsy because they require surgery for their condition. Because the research objective is to obtain specimens for neuroscience research, only participants who require a surgical procedure that requires a craniotomy and removal of brain tissue will be included.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2001-10-10 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Sample Collection | Baseline
  The goal of this protocol is to distribute human brain tissue samples to NINDS labs and collaborators.

CONTACTS AND LOCATIONS:
Overall Officials: Kareem A Zaghloul, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ojemann GA. Temporal lobe epilepsy. Clin Neurosurg. 1997;44:79-90. No abstract available. PMID 10080003
- [Background] Sperling MR, Feldman H, Kinman J, Liporace JD, O'Connor MJ. Seizure control and mortality in epilepsy. Ann Neurol. 1999 Jul;46(1):45-50. doi: 10.1002/1531-8249(199907)46:13.0.co;2-i. PMID 10401779
- [Background] Yasargil MG, Wieser HG, Valavanis A, von Ammon K, Roth P. Surgery and results of selective amygdala-hippocampectomy in one hundred patients with nonlesional limbic epilepsy. Neurosurg Clin N Am. 1993 Apr;4(2):243-61. No abstract available. PMID 8467211
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-N-0014.html